CLINICAL TRIAL: NCT00000805
Title: A Pharmacokinetic and Tolerance Study of Oral Ganciclovir in HIV-Infected Children With Asymptomatic Cytomegalovirus Infection and Low CD4 Cell Counts or Quiescent Cytomegalovirus Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 226; 11203 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Cytomegalovirus Infections; HIV Infections
Keywords: Ganciclovir; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Cytomegalovirus Infections; HIV Infections; Multiple Acyl Coenzyme A Dehydrogenase Deficiency; Acquired Immunodeficiency Syndrome | interventions — Ganciclovir

INTERVENTIONS:
Drug: Ganciclovir

SUMMARY:
PRIMARY: To determine the pharmacokinetics, MTD, and long-term safety and tolerance of oral ganciclovir in HIV-infected infants, children, and adolescents.

SECONDARY: To evaluate the effect of oral ganciclovir on the virologic parameters of CMV.

Maintenance treatment with intravenous (IV) ganciclovir for cytomegalovirus retinitis in AIDS patients is now standard therapy, but daily IV therapy can be complicated by catheter infections and thrombosis. An oral regimen of ganciclovir has been administered safely in adult AIDS patients and may be of significant benefit to children and infants as well.

DETAILED DESCRIPTION:
Maintenance treatment with intravenous (IV) ganciclovir for cytomegalovirus retinitis in AIDS patients is now standard therapy, but daily IV therapy can be complicated by catheter infections and thrombosis. An oral regimen of ganciclovir has been administered safely in adult AIDS patients and may be of significant benefit to children and infants as well.

Patients are assigned to 1 of 5 (PER AMENDMENT 10/24/95, was 4) oral (syrup or capsules) dose levels following a single intravenous dose of ganciclovir. Treatment continues for 72 (PER AMENDMENT 10/24/95, was 24 weeks) weeks after the last patient has been enrolled.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

PER AMENDMENT 10/24/95: Allowed:

* All antiretroviral agents and other medications except those listed under Exclusion - Concurrent Medications.
* Didanosine. However, patients receiving both drugs (didanosine and ganciclovir) should be monitored for toxicity.
* Amphotericin B is allowed but requires additional monitoring.

Patients must have:

* HIV infection.
* CMV infection.
* CD4 count < 150 cells/mm3 or < 15 percent AND/OR quiescent CMV disease.
* NO loss of sight from CMV retinitis.
* NO acute opportunistic infection.
* Life expectancy at least to study completion.
* Consent of parent or guardian.

NOTE:

* Infants < 6 months of age at enrollment must have been >= 36 weeks gestational age at birth.

NOTE:

* Patients may co-enroll in other ACTG protocols that do not involve the administration of disallowed medications.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Loss of sight in one eye for any reason, with evidence of CMV retinitis in the other eye.
* Acute or chronic diarrhea that would affect absorption.
* Clinical or laboratory toxicities of grade 3 or worse.

Concurrent Medication:

Excluded:

* Foscarnet.
* Acyclovir.
* Interferon.
* Myelotoxic agents for malignancy or other condition.
* Other agents with anti-CMV activity. (NOTE:

Enrollment of patients on IVIG must be discussed with protocol chair.)

* Imipenem/cilastatin sodium.

Prior Medication:

Excluded within 30 days prior to study entry:

* G-CSF or GM-CSF.

Ages: 14 Days to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32
Dates: Study Completion 1998-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frenkel L, Study Chair; Dankner W, Study Chair
Locations (19):
- United States (18):
  - Childrens Hosp. LA - Dept. of Ped., Div. of Clinical Immunology & Allergy, Los Angeles, California
  - Usc La Nichd Crs, Los Angeles, California
  - UCLA-Los Angeles/Brazil AIDS Consortium (LABAC) CRS, Los Angeles, California
  - Children's Hosp. & Research Ctr. Oakland, Ped. Clinical Research Ctr. & Research Lab., Oakland, California
  - UCSD Maternal, Child, and Adolescent HIV CRS, San Diego, California
  - Harbor - UCLA Med. Ctr. - Dept. of Peds., Div. of Infectious Diseases, Torrance, California
  - Univ. of Colorado Denver NICHD CRS, Aurora, Colorado
  - Univ. of Miami Ped. Perinatal HIV/AIDS CRS, Miami, Florida
  - Chicago Children's CRS, Chicago, Illinois
  - Tulane/LSU Maternal/Child CRS, New Orleans, Louisiana
  - HMS - Children's Hosp. Boston, Div. of Infectious Diseases, Boston, Massachusetts
  - BMC, Div. of Ped Infectious Diseases, Boston, Massachusetts
  - St. Joseph's Hosp. & Med. Ctr. of New Jersey, Paterson, New Jersey
  - Columbia IMPAACT CRS, New York, New York
  - Incarnation Children's Ctr., New York, New York
  - NYU Med. Ctr., Dept. of Medicine, New York, New York
  - St. Christopher's Hosp. for Children, Philadelphia, Pennsylvania
  - UW School of Medicine - CHRMC, Seattle, Washington
- Univ. of Puerto Rico Ped. HIV/AIDS Research Program CRS, San Juan, Puerto Rico

REFERENCES:
- [Background] Capparelli EV, Frenkel LM, Dankner W, Wei LJ, Xu J, Spector S, Connor J, Ballow A, Mohan K, Robinson C, Shaver A, Rich K, Thompson M, Read J, Wirkus C, Balsley J, Culnane M, Mcintosh K. Population pharmacokinetics of oral and intravenous ganciclovir (GCV) in HIV and CMV infected children. Program Abstr Intersci Conf Antimicrob Agents Chemother. 1996 Sep 15-18:10 (abstract no A51)
- [Background] Frenkel LM, Dankner W, Capparelli E, Wei LJ, Xu J, Spector S, Connor J, Ballow A, Mohan K, Robinson C, Shaver A, Rich K, Thompson M, Read J, Wirkus C, Balsley J, Culnane M, McIntosh K. A pharmacokinetic (PK) study of oral ganciclovir (GCV) in HIV- and cytomegalovirus (CMV)- infected children. Int Conf AIDS. 1996 Jul 7-12;11(2):31 (abstract no WeB550)
- [Background] Frenkel LM, Capparelli EV, Dankner WM, Xu J, Smith IL, Ballow A, Culnane M, Read JS, Thompson M, Mohan KM, Shaver A, Robinson CA, Stempien MJ, Burchett SK, Melvin AJ, Borkowsky W, Petru A, Kovacs A, Yogev R, Goldsmith J, McFarland EJ, Spector SA. Oral ganciclovir in children: pharmacokinetics, safety, tolerance, and antiviral effects. The Pediatric AIDS Clinical Trials Group. J Infect Dis. 2000 Dec;182(6):1616-24. doi: 10.1086/317600. Epub 2000 Nov 8. PMID 11069232